CLINICAL TRIAL: NCT04348201
Title: Foot Reflexology Combined With Dietary Modification on Premenstrual Syndrome
Brief Title: Foot Reflexology on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo Un 89
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Reflexology; Dietary Modification
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Fifty volunteer, single females with premenstrual syndrome (PMS) were selected randomly from outpatient clinic of obstetrics and gynecology at Kasr El Ainy University Hospital, Faculty of Medicine, Cairo University to share in this study, their age ranged from 18 to 25 years old and their body mass index (BMI) did not exceed 30kg/m2, the participants were assigned into two groups of equal numbers. The group (A) received therapeutic foot reflexology with dietary modification 3 times/week for8 weeks, while the group (B) received dietary modifications only for 8 weeks
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology (Active Comparator): foot reflexology session which takes about 20 minutes.
  Interventions: Other: foot reflexology
- dietary modification (Active Comparator): diet must be rich in vitamins.
  Interventions: Dietary Supplement: dietary modification

INTERVENTIONS:
Other: foot reflexology — foot reflexology session which takes about 20 minutes. The position of the patient during reflexology session was a relaxed comfortable supine lying position. The therapist was sitting position at the level of the feet. The Session of reflexology was done on three points at both feet.
  Arms: foot reflexology
Dietary Supplement: dietary modification — diet must be rich in vitamins as fish and beans, calcium as milk and chess, low fat food through decrease oil in meals, high fiber food through all types of vegetables and fruits and restrict caffeine
  Arms: dietary modification

SUMMARY:
: Premenstrual Syndrome (PMS) is a set of physical, emotional and behavioral symptom that start during the week preceding menstruation and are alleviated when the menstrual flow begins. Reflexology is one of the most popular complementary therapies

DETAILED DESCRIPTION:
This study was aimed to determine the effect of foot reflexology in the treatment of premenstrual syndrome. Subjects and methods: Fifty volunteer, single females with premenstrual syndrome (PMS) were selected randomly from outpatient clinic of obstetrics and gynecology at Kasr El Ainy University Hospital, Faculty of Medicine, Cairo University to share in this study, their age ranged from 18 to 25 years old and their body mass index (BMI) did not exceed 30kg/m2, the participants were assigned into two groups of equal numbers. The group (A) received therapeutic foot reflexology with dietary modification 3 times/week for8 weeks, while the group (B) received dietary modifications only for 8 weeks. All subjects in both groups were assessed through the visual analogue scale (VAS) for pain and Premenstrual Daily Symptoms Questionnaire for (PMS) related symptoms. Results: The results of the present study revealed that there was statistically significant improvement in both pain and premenstrual related symptoms in group (A) than in group (B).

ELIGIBILITY:
Inclusion Criteria:

* their age ranged from 18 to 25 years old
* their body mass index (BMI) did not exceed 30kg/m2

Exclusion Criteria:

* Rheumatoid arthritis
* Bronchial asthma
* depression
* anxiety

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 8 weeks
  was used to measure the severity of pain for each female in both groups (A, B) before and after the treatment according to 5 cm calibrated line with 0 (zero) representing no pain and 5 representing worst pain, each female in both groups (A&B) would be asked to mark on the line that represents her level of pain before and after treatment.

SECONDARY OUTCOMES:
Premenstrual daily symptoms questionnaire | 8 weeks
  were taken for all participants in both groups (A&B) through asked all patients all questions in the questionnaire by: were you have symptoms such as: tension, anger, anxiety, depression and crying